CLINICAL TRIAL: NCT01753024
Title: The Incidence of Pancreatic Exocrine Insufficiency and the Benefits of Pancreatic Enzyme Supplementation in Critically Ill Adult Patients
Brief Title: Pancreatic Exocrine Insufficiency and Pancreatic Enzyme Supplementation in Critically Ill Adult Patients
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Tongji Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Sheng Wang MD PhD, Associate professor, Shanghai 10th People's Hospital
Other Study IDs: STPH-ICU-001
Record Dates: First submitted 2012-12-16; First posted 2012-12-20 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Critical Illness; Sepsis; Diabetes; Cardiac Arrest; Acute Renal Failure; Shock
Keywords: exocrine pancreatic insufficiency; fecal elastase-1; amylase; lipase; critical illness; enteral nutrition; malnutrition; sepsis; diabetes; hyperlactacidemia; hemodialysis; mechanical ventilation
MeSH Terms: conditions — Critical Illness; Sepsis; Diabetes Mellitus; Heart Arrest; Acute Kidney Injury; Shock; Exocrine Pancreatic Insufficiency; Malnutrition; Hyperlactatemia | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples: lactate, hemoglobin, total bilirubin, trypsin, Vit D, etc. Stool samples: 24h fecal fat; fetal elastase-1; Fecal chymotrypsin. Nutrition status: BMI, weight loss, biomarkers such as albumin and prealbumin, etc.
  Radiological assessments: MRCP & CT scanning.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Sepsis-PEST: septic patients with enteral nutrition and pancreatic enzyme supplementation therapy
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- Sepsis-NPEST: Septic patients with enteral nutrition only
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- DM-PEST: Diabetic patients with enteral nutrition and pancreatic enzyme supplementation therapy
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- DM-NPEST: Diabetic patients with enteral nutrition only
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- PCAS-PEST: Patients suffering from cardiac arrest receive both enteral nutrition and pancreatic enzyme supplementation therapy
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- PCAS-NPEST: Patients suffering from cardiac arrest receive enteral nutrition only
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- ARF-PEST: Patients with acute renal failure receive both enteral nutrition and pancreatic enzyme supplementation therapy
  Interventions: Dietary Supplement: Enteral nutrition (EN)
- ARF-NPEST: Patients with acute renal failure receive enteral nutrition only
  Interventions: Dietary Supplement: Enteral nutrition (EN)

INTERVENTIONS:
Dietary Supplement: Enteral nutrition (EN) — All patients enrolled in this study must carry out nutritional support by enteral nutrition

SUMMARY:
Malnutrition is a frequent problem in critically ill patients that is associated with detrimental clinical outcomes. To provide adequate nutritional support, current studies focused mostly on the choice of delivery timing, formula selection and the route of administration, little attention was paid to malnutrition related to exocrine pancreatic insufficiency (EPI).

In fact, malnutrition is also a major consequence of pancreatic exocrine insufficiency and pancreatic damage is commonly observed in critically ill patients without prior pancreatic diseases. Hence, EPI associated malnutrition should be concerned due to the high prevalence of pancreatic damage in critically ill patients.

The aims of this study is to evaluate the incidence of EPI in critically ill adult patients and explore its potential risk factors. Moreover, the efficacy of pancreatic enzyme supplementation therapy on malnutrition in ICU patients with specific clinical characteristics will be investigated.

DETAILED DESCRIPTION:
Critically ill patients who is able to receive early enteral nutrition and estimated to stay in ICU at least four days are considered to enroll into this study. Exclusion criteria are age under 18 or over 80 years, pregnancy or breastfeeding, known exocrine pancreatic insufficiency due to pancreatitis, unresectable pancreatic cancer, cystic fibrosis, celiac disease, Zollinger-Ellison syndrome, pancreatectomy, gastrectomy and medications of somatostatin or aprotinin that directly influence pancreatic exocrine function.

Informed consent documents are signed by immediate family members of the recruited patients. All study procedures are performed in accordance with the institutional guidelines for the conduct of research on human beings and approved by the Human Ethics Committee of Shanghai Tenth People's Hospital.

Once the enrolled patients are admitted to the ICU, they are inserted either a nasogastric tube or a nasojejunal tube guided by electronic gastroscope according to the expected feeding time, and the position of feeding tubes is confirmed by plain abdominal radiograph. Enteral nutrition will be initiated at a rate of 25 ml/h within 24h of admission, and the infusion rate increases steadily until the prescribed nutritional requirements are achieved within 3 days. Daily nutritional requirements are calculated mainly based on the patient's body mass index.

During the study, the details of each patient such as age, sex, BMI, admission diagnosis, and Acute Physiology and Chronic Health Evaluation II score are collected. All clinical characteristics that may cause pancreatic damage, including shock (systolic blood pressure < 90 mmHg), tissue hypoxia (serum lactate > 2 mmol/L), respiratory failure (PaO2 < 60 mmHg), anemia (hemoglobin < 90 g/L), obesity (BMI > 30 kg/m2), biliary sludge (total bilirubin > 17.5 μmol/L), hypertriglyceridemia (> 1.7 mmol/L), sepsis, cardiac arrest, cardiopulmonary bypass (CPB), severe head injury, acute stroke, post-neurosurgery, diabetes, inflammatory bowel disease (IBS), mechanical ventilation and continuous renal replacement therapy (CRRT) are recorded prospectively. Medications such as propofol, valproate, metronidazole and morphine-derived drugs, which are applied for more than 24 h and might induce pancreatic damage, are also documented. Arterial blood samples are taken 3 days after admission to determine biochemical parameters. Stool samples are collected 3-5 days after the beginning of enteral nutrition and frozen at -20℃ until analysis. Some patients will undergo CT scanning and magnetic resonance cholangio-pancreatography (MRCP)to acquire histological evidence of exocrine pancreatic insufficiency.

ELIGIBILITY:
Inclusion Criteria: All critically ill patients who are able to receive early enteral nutrition and estimated to stay in ICU at least four days

Exclusion Criteria: age under 18 or over 80 years, pregnancy or breastfeeding, known exocrine pancreatic insufficiency due to pancreatitis, unresectable pancreatic cancer, cystic fibrosis, celiac disease, Zollinger-Ellison syndrome, pancreatectomy, gastrectomy and medications of somatostatin or aprotinin that directly influence pancreatic exocrine function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill patients who are able to receive early enteral nutrition and estimated to stay in ICU at least four days
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Screening and risk factors of exocrine pancreatic insufficiency in critically ill adult patients receiving enteral nutrition | From 2012-1 to 2012-12
  The incidence of exocrine pancreatic insufficiency will be evaluated that is based on hyperamylasemia, hyperlipasemia and fecal elastase-1 concentrations. multivariate logistic regression analyses are used to estimate the correlations between exocrine pancreatic insufficiency and clinical events and characteristics, which include APACHE II score, shock, hyperlactacidemia, respiratory failure, anemia, obesity, biliary sludge, hypertriglyceridemia, sepsis, cardiac arrest, cardiopulmonary bypass, severe head injury, acute stroke, post-neurosurgery, diabetes, inflammatory bowel disease, mechanical ventilation, continuous renal replacement therapy and medications such as propofol, valproate, metronidazole and morphine-derived drugs

SECONDARY OUTCOMES:
Effects of pancreatic enzyme supplementation on nutritional status and clinical outcomes in critically ill patients with sepsis | From 2013-1 to 2014-12
  The incidence of exocrine pancreatic insufficiency and the nutritional status are evaluated by fecal elastase-1 concentrations before pancreatic enzyme supplementation therapy is applied.
  Patients are assigned into two groups randomly, the control group is only receiving enteral nutrition without the addition of pancreatic enzyme(CREON), and the PEST group is given both enteral nutrition and pancreatic enzyme supplementation therapy at the same time.
  Following two weeks of corresponding treatments, the nutritional status and clinical outcomes are documented in both groups for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Wang, MD, PhD, Study Director — Shanghai 10th People's Hospital; Yu G Zhuang, MD, MSc, Principal Investigator — Shanghai 10th People's Hospital; Li J Ma, MD, MSc, Principal Investigator — Shanghai 10th People's Hospital
Locations (2):
- China (2):
  - Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Larger E, Philippe MF, Barbot-Trystram L, Radu A, Rotariu M, Nobecourt E, Boitard C. Pancreatic exocrine function in patients with diabetes. Diabet Med. 2012 Aug;29(8):1047-54. doi: 10.1111/j.1464-5491.2012.03597.x. PMID 22273174
- [Background] Teichmann J, Riemann JF, Lange U. Prevalence of exocrine pancreatic insufficiency in women with obesity syndrome: assessment by pancreatic fecal elastase 1. ISRN Gastroenterol. 2011;2011:951686. doi: 10.5402/2011/951686. Epub 2011 Nov 3. PMID 22111014
- [Background] Wier HA, Kuhn RJ. Pancreatic enzyme supplementation. Curr Opin Pediatr. 2011 Oct;23(5):541-4. doi: 10.1097/MOP.0b013e32834a1b33. PMID 21799412
- [Background] Leeds JS, Oppong K, Sanders DS. The role of fecal elastase-1 in detecting exocrine pancreatic disease. Nat Rev Gastroenterol Hepatol. 2011 May 31;8(7):405-15. doi: 10.1038/nrgastro.2011.91. PMID 21629239
- [Background] Ferrie S, Graham C, Hoyle M. Pancreatic enzyme supplementation for patients receiving enteral feeds. Nutr Clin Pract. 2011 Jun;26(3):349-51. doi: 10.1177/0884533611405537. Epub 2011 Apr 20. PMID 21508176
- [Background] Dominguez-Munoz JE. Pancreatic exocrine insufficiency: diagnosis and treatment. J Gastroenterol Hepatol. 2011 Mar;26 Suppl 2:12-6. doi: 10.1111/j.1440-1746.2010.06600.x. PMID 21323992
- [Background] Kuhn RJ, Gelrud A, Munck A, Caras S. CREON (Pancrelipase Delayed-Release Capsules) for the treatment of exocrine pancreatic insufficiency. Adv Ther. 2010 Dec;27(12):895-916. doi: 10.1007/s12325-010-0085-7. Epub 2010 Nov 15. PMID 21086085
- [Background] Griesche-Philippi J, Otto J, Schworer H, Maisonneuve P, Lankisch PG. Exocrine pancreatic function in patients with end-stage renal disease. Clin Nephrol. 2010 Dec;74(6):457-64. doi: 10.5414/cnp74457. PMID 21084049
- [Background] Ockenga J. Importance of nutritional management in diseases with exocrine pancreatic insufficiency. HPB (Oxford). 2009 Dec;11 Suppl 3(Suppl 3):11-5. doi: 10.1111/j.1477-2574.2009.00134.x. PMID 20495627
- [Background] Hardt PD, Mayer K, Ewald N. Exocrine pancreatic involvement in critically ill patients. Curr Opin Clin Nutr Metab Care. 2009 Mar;12(2):168-74. doi: 10.1097/MCO.0b013e328322437e. PMID 19202388
- [Background] Senkal M, Ceylan B, Deska T, Marpe B, Geier B. Exocrine pancreas disfunction in severely traumatised patients and early enteral nutrition. Ulus Travma Acil Cerrahi Derg. 2008 Jan;14(1):34-9. PMID 18306065
- [Background] Denz C, Siegel L, Lehmann KJ, Dagorn JC, Fiedler F. Is hyperlipasemia in critically ill patients of clinical importance? An observational CT study. Intensive Care Med. 2007 Sep;33(9):1633-6. doi: 10.1007/s00134-007-0668-1. Epub 2007 May 12. PMID 17497124
- [Background] Nys M, Venneman I, Deby-Dupont G, Preiser JC, Vanbelle S, Albert A, Camus G, Damas P, Larbuisson R, Lamy M. Pancreatic cellular injury after cardiac surgery with cardiopulmonary bypass: frequency, time course and risk factors. Shock. 2007 May;27(5):474-81. doi: 10.1097/shk.0b013e31802b65f8. PMID 17438451
- [Background] Serrano N. Increased lipase plasma levels in ICU patients: when are they critical? Chest. 2005 Jan;127(1):7-10. doi: 10.1378/chest.127.1.7. No abstract available. PMID 15653954
- [Derived] Wang S, Ma L, Zhuang Y, Jiang B, Zhang X. Screening and risk factors of exocrine pancreatic insufficiency in critically ill adult patients receiving enteral nutrition. Crit Care. 2013 Aug 7;17(4):R171. doi: 10.1186/cc12850. PMID 23924602